CLINICAL TRIAL: NCT02531074
Title: Swipe Out Stroke (SOS): Feasibility of Using a Consumer Based Electronic Application to Improve Compliance With Weight Loss in Obese Minority Stroke Patients
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nneka Lotea Ifejika, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-13-0608
Record Dates: First submitted 2015-08-20; First posted 2015-08-21 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Stroke
Keywords: Mobile Applications
MeSH Terms: conditions — Stroke

ARMS (2):
- Mobile Application plus Usual Care (Experimental)
  Interventions: Behavioral: Mobile Application; Behavioral: Usual Care
- Food Journal plus Usual Care (Active Comparator)
  Interventions: Behavioral: Food Journal; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Mobile Application
  Arms: Mobile Application plus Usual Care
Behavioral: Food Journal
  Arms: Food Journal plus Usual Care
Behavioral: Usual Care

SUMMARY:
This pilot study evaluates the use of a mobile application to improve weight loss in obese stroke patients. The investigators hypothesize that acute stroke patients who use the mobile application are more likely to achieve a minimum 5% weight reduction during the critical six months post-stroke, yielding considerable improvement in stroke risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or hemorrhagic stroke.
2. Age 18-85 years.
3. African-American or Hispanic.
4. Modified Rankin Scale (mRS) of 0-3.
5. Body Mass Index greater than 30 kg/m2.
6. Currently taking prescription medication for diabetes mellitus, hypertension or hyperlipidemia.
7. Willing to follow a healthy eating pattern and NOT use weight loss medications for the duration of the study.
8. Personal ownership or caregiver ownership of a personal computer, SmartPhone or other SmartDevice (iPhone or Android platform) with Internet access.
9. If patient has alexia, agraphia, acalculia, dementia or blindness - caregiver must be willing to complete the intervention.

Exclusion Criteria:

1. Pre-existing disability with mRS > 4.
2. Contraindications to weight loss (planning to become pregnant, history of an eating disorder).
3. Steroid use for suspected vasculitis.
4. Current or recent (past 6 months) participation in a weight loss program or use of weight loss medication.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with five percent or greater weight loss. | Six months

SECONDARY OUTCOMES:
Percentage of patients with blood pressure reduction. | Six months
Percentage of patients with decrease in serum cholesterol. | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at Houston Medical School, Houston, Texas, United States

REFERENCES:
- [Result] Ifejika NL, Noser EA, Grotta JC, Savitz SI. Swipe out Stroke: Feasibility and efficacy of using a smart-phone based mobile application to improve compliance with weight loss in obese minority stroke patients and their carers. Int J Stroke. 2016 Jul;11(5):593-603. doi: 10.1177/1747493016631557. Epub 2016 Mar 8. PMID 26956032
- [Result] Ifejika NL, Bhadane M, Cai C, Noser EA, Savitz SI. Cluster Enrollment: A Screening Tool for Stroke Risk Factors in Minority Women Caregivers. J Natl Med Assoc. 2019 Jun;111(3):281-284. doi: 10.1016/j.jnma.2018.10.013. Epub 2018 Nov 12. PMID 30442422
- [Result] Ifejika NL, Bhadane M, Cai CC, Noser EA, Grotta JC, Savitz SI. Use of a Smartphone-Based Mobile App for Weight Management in Obese Minority Stroke Survivors: Pilot Randomized Controlled Trial With Open Blinded End Point. JMIR Mhealth Uhealth. 2020 Apr 22;8(4):e17816. doi: 10.2196/17816. PMID 32319963